CLINICAL TRIAL: NCT01506336
Title: A Prospective, Multicenter, Randomized, Open-label, Active Controlled, 2-parallel Group, Phase II Study to Compare Efficacy and Safety of Masitinib at 12 mg/kg/Day to Sunitinib at 50 mg/Day in Treatment of Patients With Gastro-intestinal Stromal Tumor Resistant to Imatinib
Brief Title: Masitinib in Patients With Gastro-Intestinal Stromal Tumour Resistant to Imatinib
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AB Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AB07001
Record Dates: First submitted 2012-01-03; First posted 2012-01-10 (Estimated); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Gastro Intestinal Stromal Tumor
Keywords: GIST; resistant; imatinib; gastro intestinal stromal tumor resistant to imatinib
MeSH Terms: interventions — masitinib; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- masitinib (Experimental): masitinib 12 mg/kg/day
  Interventions: Drug: masitinib
- sunitinib (Active Comparator): sunitinib 50 mg/day
  Interventions: Drug: sunitinib

INTERVENTIONS:
Drug: masitinib — masitinib 12 mg/kg/day
  Arms: masitinib
Drug: sunitinib — sunitinib 50 mg/day
  Arms: sunitinib

SUMMARY:
The objective is to compare efficacy and safety of masitinib at 12 mg/kg/day to sunitinib at 50 mg/day in treatment of patients with gastro-intestinal stromal tumor resistant to imatinib.

ELIGIBILITY:
Inclusion Criteria:

1. Histological proven, metastatic, or locally advanced and non-operable GIST
2. Measurable tumor lesions with longest diameter ≥ 20 mm using conventional techniques or ≥ 10 mm with spiral CT scan according RECIST criteria
3. C-kit (CD117) positive tumors detected immuno-histochemically and documented mutation of c-kit at any time if available
4. Patients resistant to imatinib at dose of 400 mg/day

Exclusion Criteria:

1. Patient treated for a cancer other than GIST cancer within 5 years before enrolment, with the exception of basal cell carcinoma or cervical cancer in situ
2. Patient with active central nervous system (CNS) metastasis or with history of CNS metastasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2008-10; Primary Completion 2011-09 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
overall progression free survival | up to 36 weeks
  From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 weeks

SECONDARY OUTCOMES:
overall survival | up to 36 weeks
  From date of randomization until the date of death from any cause, assessed up to 36 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Axel Le Cesne, MD, Principal Investigator — Institut Gustave Roussy, Villejuif, France
Locations (1):
- Institute Gustave Roussy (IGR), Villejuif, France

REFERENCES:
- [Result] Adenis A, Blay JY, Bui-Nguyen B, Bouche O, Bertucci F, Isambert N, Bompas E, Chaigneau L, Domont J, Ray-Coquard I, Blesius A, Van Tine BA, Bulusu VR, Dubreuil P, Mansfield CD, Acin Y, Moussy A, Hermine O, Le Cesne A. Masitinib in advanced gastrointestinal stromal tumor (GIST) after failure of imatinib: a randomized controlled open-label trial. Ann Oncol. 2014 Sep;25(9):1762-1769. doi: 10.1093/annonc/mdu237. Epub 2014 Jul 25. PMID 25122671
- See also: Publication of clinical study results — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4143095/